CLINICAL TRIAL: NCT05573126
Title: A Modular, Open-Label, Multi-Centre Phase 1/2 Dose-Finding, Optimisation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of EP0062 as Monotherapy and in Combination in Patients With Relapsed Locally Advanced or Metastatic AR+/HER-2-/ER+ Breast Cancer
Brief Title: Phase 1/2 Study to Evaluate Vosilasarm (EP0062) as Monotherapy and in Combination in Patients With Advanced or Metastatic AR+/HER-2-/ER+ Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ellipses Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EP0062-101
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hormone Receptor-positive Breast Cancer; Hormone Receptor Positive HER-2 Negative Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Module A - Vosilasarm Dose Finding (Experimental): Patients are assigned to dose level cohorts to identify optimal dose and assess safety, tolerability and PK profile.
  Interventions: Drug: Vosilasarm
- Module B - Vosilasarm+ standard of care targeted therapy (elacestrant). (Experimental): 3-6 patients enrolled, with possible expansion up to 25 patients.
  Interventions: Drug: Vosilasarm; Drug: Elacestrant
- Module B - Vosilasarm+ standard of care targeted therapy (everolimus) (Experimental): 3-6 patients enrolled, with possible expansion up to 25 patients.
  Interventions: Drug: Vosilasarm; Drug: Everolimus

INTERVENTIONS:
Drug: Vosilasarm — Vosilasarm is an orally administered investigational selective androgen receptor modulator (SARM)
  Other Names: EP0062
Drug: Elacestrant — Oral SERD
  Arms: Module B - Vosilasarm+ standard of care targeted therapy (elacestrant).
Drug: Everolimus — mTOR Inhibitor
  Arms: Module B - Vosilasarm+ standard of care targeted therapy (everolimus)

SUMMARY:
The aim of this study is to identify the optimal dose for Vosilasarm (EP0062) as monotherapy and in combination with standard-of-care therapies to assess its Safety, Tolerability, Pharmacokinetics, and Efficacy in Patients with Relapsed Locally Advanced or Metastatic AR+/HER-2-/ER+ Breast Cancer

DETAILED DESCRIPTION:
Vosilasarm (EP0062) is being investigated in this modular, interventional, open label, Phase 1/2 dose finding, optimisation and expansion study to determine the optimal dose of Vosilasarm given as monotherapy and for evaluation in combination with standard-of-care therapies in patients with Relapsed Locally Advanced or Metastatic AR+/HER-2-/ER+ Breast Cancer. Module A (phase 1 dose finding) has completed and an optimal dose has been selected for module B (phase 2 expansion).

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years or older at the time of informed consent
2. Histologically proven diagnosis of breast cancer with evidence of metastatic or locally advanced breast adenocarcinoma as defined by the American Joint Committee on Cancer/Union for International Cancer Control/Tumour Node Metastases (AJCC/UICC TNM) staging classification (8th Ed, 2017) and where no conventional therapy is available or considered appropriate by the Investigator or is declined by the patient
3. Availability of archival tumour sample (formalin-fixed, paraffin-embedded block(s) or slides from a primary tumour or biopsy of a metastatic tumour lesion or lesions); in the absence of an archival tumour sample, or if only archival bone tissue is available, a fresh biopsy will need to be collected
4. Biopsy-proven AR+ and ER+ breast cancer

   * For Module A, AR+ breast cancer is defined as ≥ 10% AR nuclei staining by central immunohistochemistry (IHC) using the Ventana assay
   * For Modules B and C, AR+ breast cancer is defined as ≥ 30% AR nuclei staining by central IHC using the Ventana assay
5. HER2-negative breast cancer, defined as negative by fluorescence in situ hybridisation (FISH) or IHC score of 0 or 1+. If IHC is equivocal at 2+, a negative FISH test (HER2/Amplification of the centromeric region of chromosome 17)CEP17 ratio of <2.0) is required
6. Postmenopausal, as defined by at least one of the following:

   1. Age over 60 years
   2. Amenorrhea > 12 months at the time of informed consent and an intact uterus, with follicle-stimulating hormone (FSH) and oestradiol in the postmenopausal ranges (as per local practice)
   3. FSH and oestradiol in the postmenopausal ranges (as per local practice) in women aged <55 years who have undergone hysterectomy
   4. Prior bilateral oophorectomy
7. Module B arm 1: patients who have progressed on ≤ 2 prior lines of endocrine therapy, including a prior CDK4/6 inhibitor.
8. Module B arm 2: patients who have progressed on ≤ 2 prior lines of endocrine therapy in advanced/metastatic setting, including prior CDK4/6 inhibitor

Exclusion Criteria:

Patients with any of the following will not be included in the study:

1. Prior anti-cancer or investigational drug treatment within the following time windows:

   * Any chemotherapy within 21 days prior to the first dose of study drug
   * Any non-chemotherapy investigational anti-cancer drug < 5 half-lives (28 days for biologics) or < 14 days for small-molecule therapeutics or if half-life is not known
   * Tamoxifen and aromatase inhibitors within 14 days prior to the first dose of study drug
   * Fulvestrant or other investigational Selective Estrogen Receptor Degraders (SERDs) within 21 days prior to first dose of study drug
2. Currently taking testosterone, methyltestosterone, oxandrolone, oxymetholone, danazol, fluoxymesterone, testosterone-like agents (e.g., dehydroepiandrosterone, androstenedione, and other androgenic compounds, including herbals), or antiandrogens
3. Radiation therapy within 14 days prior to the first dose of study drug and scheduled to have radiation therapy during participation in this study. Short courses of palliative radiation therapy during the study might be allowed following discussion with and approval by the Medical Monitor. Palliative radiotherapy within 6 weeks prior to first dose of study drug is permitted
4. Unresolved or unstable serious toxic side effects of prior chemotherapy or radiotherapy, i.e., ≥ Grade 2 per Common Terminology Criteria for Adverse Events (CTCAE) v5.0, except fatigue, alopecia, and Grade 2 chemotherapy-induced neuropathy
5. Confirmed Corrected QT Interval by Fridericia (QTcF) > 470 ms on screening ECG, or history of torsades de pointes (TdP), or history of congenital long QT syndrome, or immediate family history of long QT syndrome, unexplained sudden death at a young age, or sudden cardiac death
6. Any other clinically important abnormalities in rhythm, conduction, or morphology on resting ECG (e.g., complete left bundle branch block, third-degree heart block); rate-controlled atrial fibrillation is permitted
7. Concomitant medications that prolong the corrected QT interval and/or increase the risk for TdP that cannot be discontinued or substituted with another drug within 5 half-lives or 14 days before the first dose of study drug, whichever is longer
8. Congestive heart failure Grades II-IV according to the New York Heart Association at the time of screening
9. Myocardial infarction or unstable angina within the previous 6 months
10. Patients receiving medications that are known to be strong inhibitors or inducers of CYP3A4 within 5 half-lives or 14 days, whichever is longer, before the first dose of study drug
11. Prior treatment with selected combination agent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) during Cycle 1 of EP0062 treatment | first 28 days
  Module A
Maximum tolerated dose (MTD) and doses for evaluation in the expansion cohorts | 1 year
  Module A
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | up to 30 days after the end of treatment
  Module A/B
Recommended clinical (dose (s) for combination therapy | 1 year
  Module B

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters - Half life | 1, 2, 4, 8, 24 and 48 hours during cycle 1
Plasma pharmacokinetic (PK) parameters - Cmax | 1, 2, 4, 8, 24 and 48 hours during cycle 1
Plasma pharmacokinetic (PK) parameters - Area under the curve (exposure) | 1, 2, 4, 8, 24 and 48 hours during cycle 1
Tumour response | screening and every 8 weeks up to 12 months
Clinical Benefit Rate (CBR) | every 8 weeks up to 12 months
Objective Response Rate (ORR) | every 8 weeks up to 12 months
Duration of Response (DOR) | every 8 weeks up to 12 months
Progression-free survival (PFS) | every 8 weeks up to 12 months
Overall Survival (OS) | every 8 weeks up to 12 months
Relationship between EP0062 efficacy parameters and the level of Androgen Receptor expression and Androgen Receptor : Oestrogen Receptor ratio | every 8 weeks up to 12 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (7):
  - Yale School of Medicine, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology Baylor University Medical Center, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Spain (4):
  - Hospital 12 de Octubre, Usera, Madrid
  - Hospital Universitari Vall d'Hebron (VHIO), Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - NEXT Oncology Hospital Quironsalud, Madrid
- United Kingdom (3):
  - Sarah Cannon Research Institute UK, London, Harley Saint
  - The Christie NHS Foundation Trust, Manchester, Wilmslow Rd
  - The Clatterbridge Cancer Centre, Liverpool